CLINICAL TRIAL: NCT05905185
Title: Interventional Strategy in Tackling Emerging Non-alcoholic Fatty Liver Disease in Childhood Obesity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GUP 2018-052
Record Dates: First submitted 2023-05-01; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Obesity
Keywords: obesity; Non-alcoholic Fatty Liver Disease; Children; Tocotrienol-Rich Fraction Vitamin E
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Sime Darby Bioganic Sdn. Bhd, Malaysia provided the TRF pills that were used in the study. The 50 mg of vitamin E isomers in the TRF included 17.1 mg of α-tocopherol ,18.28 mg of α- tocotrienol, 2.02 mg of β-tocotrienol, 22.3 mg of γ-tocotrienol and 7.4 mg of δ-tocotrienol. During a period of six months, the patients were instructed to consume oral TRF (50 mg) daily
  Interventions: Drug: Tocotrienol-rich fraction vitamin E (TRF)
- Placebo (Placebo Comparator): During a period of six months, the patients were instructed to consume oral placebo (50 mg) pills daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tocotrienol-rich fraction vitamin E (TRF) — The 50 mg of vitamin E isomers in the TRF included 17.1 mg of α-tocopherol ,18.28 mg of α- tocotrienol, 2.02 mg of β-tocotrienol, 22.3 mg of γ-tocotrienol and 7.4 mg of δ-tocotrienol.
  Arms: Treatment
Drug: Placebo — 50mg of Placebo
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effects of tocotrienol-rich fraction vitamin E supplementation on liver enzymes in overweight and obese children with non-alcoholic fatty liver disease as compared to placebo.

The main question[s] it aims to answer are:

1. Does supplementation of tocotrienol-rich fraction vitamin E reduce the level of liver enzymes and improve liver steatosis in non-alcoholic fatty liver disease among overweight and obese children?
2. Does tocotrienol-rich fraction vitamin E supplementation improve the level of liver steatosis by reducing the level of DNA damage?

Participants will :

1. consume daily either a dose of 50 mg of tocotrienol-rich fraction (TRF) vitamin E or a placebo for 6 months.
2. Routine clinical assessments include weight, height, waist circumference, and BMI. Fasting glucose, and fasting serum lipid.
3. The following investigations were performed upon recruitment and following 6 months of intervention: (i) liver biomarker and enzymes; (ii) DNA damage; (iii) TNFα, IL-6 and IFN-gamma genes; (iv) Fibroscan.

DETAILED DESCRIPTION:
Methodology This study enrolled a diverse group of participants aged 10 to 18, regardless of gender, who were diagnosed with fatty liver disease detected via ultrasonography and abnormally high alanine transaminase levels (at least two-fold higher than the upper limits for their respective genders). The trial consisted of 29 patients, with 15 receiving a daily oral dose of 50 mg TRF and 14 receiving a placebo for a duration of six months. Various clinical parameters, LIVERFASt in vitro diagnostic test, fibroscan, biochemical parameters, DNA damage, and gene expression, both at the outset and at the end of the study were monitored.

The amount of blood sample taken was 13mls each at entry and on completion at 6 months. Details of these tests are as shown below:

Transient Elastography (FibroScan):

This is a non-invasive test to measure liver stiffness, kPa (indicator of liver fibrosis) and to detect degree of fat accumulation (CAP range value of 100-400 dB/m), liver stiffness of > 8kPa indicates advanced fibrosis while CAP of > 263 indicates fatty liver. During the screening, the participant lied down on the examination bed with his/her right hand behind his/her head. A probe was placed by the investigator between the right ribs of the patient. Measurements were recorded into the machine (FibroScan® 502 Touch). The screening is quick and easy, usually taking less than 15 minutes. The scanned steatosis was scored and graded.

Determination of DNA Damage The DNA Damage pre and post intervention were conducted by using CometAssay Kit (Trevigen, Gaithersburg, USA) following the manufacturer's protocol. Briefly, blood cells in 5 μL medium was suspended in 70 μL warm 0.6% low-melting point (LMA) agarose (Boehringer Mannheim, Germany) (DNAse-free, RNAsefree). Slides were allowed to sit in the alkaline buffer for 20 min to allow unwinding of DNA strands and expression of alkali-labile damage. Electrophoresis was performed for 20 min at 300 mA and 25 V. Following dropwise neutralization (TrisHCl, pH 7.5) for 5 min, cells were stained by applying 30 μL 1X ethidium bromide. The slides were examined and the tail length was measured with a fluorescence microscope (Carl Zeiss, Germany). The DNA migration of 100 randomly selected cells were examined for each sample. A total damage score was determined by multiplying the number of cells assigned to each grade of damage by the numeric value of the grade according to methods described by Heaton et al. [19]. Total DNA damage score was calculated as follows. Total DNA damage = [(0 × n0) + (1 × n1) + (2 × n2) + (3 × n3) + (4 × n4)] where n0 =cells with Score 0, n1 = cells with Score 1, n2 = cells with Score 2, n3 = cells with Score 3, and n4 = cells with Score 4.

Determination of liver biomarker and enzyme The levels of liver enzymes including alanine aminotransferase, ALT, aspartate aminotransferase, AST, gamma glutamyl transferase, GGT, and alkaline phosphatase, ALP, pre and post intervention were determined from the blood samples of the patients. Other biomarkers such as lipid profile, α-2 macroglobulin and haptoglobin were also be analysed. The blood samples were collected in a BD Vacutainer and centrifuge at 1500 xg for 15 mins for the serum separation. The serum was stored in -80°C if it is not processed immediately. The levels of the liver enzymes were determined by using ADVIA 1800 (Siemens, USA).

Quantitative Polymerase Chain Reaction (qPCR):

Total RNA was extracted from blood samples of NAFLD patients with or without tocotrienol. Primers and probes for TNFα, IL-6 and IFN-gamma genes were designed. 1 ug/ul of total RNA was converted to cDNA which then be used for PCR reaction. All samples were analysed in duplicate. Expression of genes was determined after normalised with the housekeeping genes.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 13 - 18 years old
2. Overweight or obese (BMI percentile range ≥ 85%)
3. Able to swallow small oral soft gel capsule
4. Diagnosis of NAFLD confirmed by presence of fatty liver detected by abdominal ultrasound and controlled attenuation parameter (CAP) score of >263
5. Elevated alanine transaminase (ALT) ≥ 2 fold upper limits (26 U/L for boys and 22 U/L for girls)

Exclusion Criteria:

* Evidence of other primary chronic liver diseases (as determined by clinical and standard investigations) - e.g. Hepatitis B, C infections, autoimmune hepatic disorders.
* Not on any dietary supplements.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Mean difference of fibrosis score, inflammation (activity) score and steatosis score | Six months
  Serum LiverFASt level is a blood test to detect the degree and stage of: fibrosis (0-1), inflammation (0-1), and steatosis (0-1) scores. The higher the score indicates the higher the degree of fibrosis, inflammation and steatosis. These measurements were taken at the baseline and at the end of trial.
Mean difference of fasting blood glucose | 6 months
  Fasting blood glucose levels were measured at the baseline and at the end of trial
Mean difference in aspartate aminotransferase & alanine aminotransferase levels | 6 months
  Aspartate aminotransferase & alanine aminotransferase levels were measured at the baseline and at the end of trial.
Mean difference in apolipoprotein-A1, triglycerides, total cholesterol levels | 6 months
  Total cholesterol, triglycerides, apolipoprotein-A1 levels were measured at the baseline and at the end of trial
Mean difference of liver steatosis and liver stiffness, measured by controlled attenuation parameter (CAP) score in percentage and kPa respectively, by transient elastography | 6 months
  Transient elastography was performed to measure controlled attenuation parameter (%) and liver stiffness (kPa) at the baseline and at the end of trial

SECONDARY OUTCOMES:
Mean difference in tail length to represent DNA damage | 6 months
  Determination of DNA damage using comet assay was done at the baseline and at the end of trial
Mean difference in the interleukin-6, TNF-alpha and interferon-gamma | 6 months
  IL-6, TNF-alpha and interferon-gamma levels were measured at the baseline and at the end of trial
Mean difference in the body mass index (percentile) | 6 months
  Weight measurement based on age was measured at the baseline and at the end of trial

CONTACTS AND LOCATIONS:
Overall Officials: Norfilza Mohd Mokhtar, Principal Investigator — National University of Malaysia
Locations (1):
- National University Of Malaysia, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Al-Baiaty FDR, Ishak S, Mohd Zaki F, Masra F, Abdul Aziz DA, Wan Md Zin WN, Yee Hing E, Kuthubul Zaman AS, Abdul Wahab N, Muhammad Nawawi KN, Hamid Z, Raja Ali RA, Mokhtar NM. Assessing the efficacy of tocotrienol-rich fraction vitamin E in obese children with non-alcoholic fatty liver disease: a single-blind, randomized clinical trial. BMC Pediatr. 2024 Aug 20;24(1):529. doi: 10.1186/s12887-024-04993-8. PMID 39160468